CLINICAL TRIAL: NCT02362542
Title: Effect of Transcranial Direct Current Stimulation (tDCS) on Appetite Control Related Brain Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungbuk National University (Other)
Responsible Party: Principal Investigator, Hyung Jin Choi, Clinical Assistant Professor, Chungbuk National University
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-02-014
Record Dates: First submitted 2015-02-02; First posted 2015-02-13 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sham tDCS (Experimental): Subjects will receive tDCS two times, one is active stimulation and the other is sham stimulation. Both stimulations will be separated at least one week and the order of sham and active tDCS will be counterbalanced across subjects.
  Interventions: Device: tDCS
- Real tDCS (Experimental): Subjects will receive tDCS two times, one is active stimulation and the other is sham stimulation. Both stimulations will be separated at least one week and the order of sham and active tDCS will be counterbalanced across subjects.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — For active tDCS, a 2 mA current will be delivered for 20 minutes with 20 second up and down ramp times. The anodal electrode will be placed on the right DLPFC (F4; 10-20 EEG system), and the cathode electrode will be placed on the left DLPFC (F4;10-20 EEG system), which is known to be related to cognitive function. The electrodes used for tDCS are saline-soaked sponges (25 cm2).

SUMMARY:
The purpose of this study is to investigate the effect of Transcranial Direct Current Stimulation (tDCS) on appetite control related brain regions.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is emerging tool for brain modulation in a variety of clinical conditions. In addition, recent neuroimaging studies suggest that modifying the activity of brain circuits involved in eating behavior could provide therapeutic benefits in obesity.

The investigators aim to assess whether modulation of the dorsolateral prefrontal cortex (DLFPC) using tDCS, modifies behavioral response and brain activity while watching visually presented food cues in obese subjects.

Subjects will receive tDCS two times, one is active stimulation and the other is sham stimulation. Both stimulations will be separated at least one week and the order of sham and active tDCS will be counterbalanced across subjects.

Subjects will perform functional MRI experiments with visual food cues. Questionnaire with behavior measures, body compositions, blood tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 28 kg/m2

Exclusion Criteria:

* history of brain trauma, epilepsy, or other neurological problems

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Regional brain activity measured by blood-oxygen-level dependent (BOLD) signal of functional MRI | Immediately after intervention
  3T MR scanner with Echo Planar Imaging(EPI) capability(Magnetom, Siemens Medical System)

SECONDARY OUTCOMES:
Behavior outcomes on the visual analog scale | Immediately after intervention
  Hunger related visual analogue scale (VAS) - 8 items (Flint et al., 2000) Mood related visual analogue scale (VAS) - 16 items (Fregni et al., 2008)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University, Cheongju-si, North Chungcheong, South Korea